CLINICAL TRIAL: NCT05215171
Title: World Trade Center Particulate Matter Induced Cardiorespiratory and Vascular Dysfunction: a MultiOmic Approach (CaRVD)
Status: Recruiting | Type: Observational
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute for Occupational Safety and Health (NIOSH/CDC) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: 21-00682
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Cardiorespiratory and Vascular Dysfunction; Obstructive Airway Disease
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- World Trade Center - Airway Hyperreactivity (WTC-AHR): WTC-AHR cases are defined as having either a positive MCT (PC20<16) and/or positive BDR (by ATS/ERS guidelines with improvement of FEV1 by 12% and at least 200mL) post-9/11.
- Control Group: Cohort Controls will be randomly selected 10% of the baseline cohort

SUMMARY:
Particulate matter (PM) associated cardiorespiratory and vascular dysfunction (CaRVD) poses a significant global health burden. The World Trade Center (WTC) destruction on September 11, 2001 led to an intense deposition of particulate matter (WTC-PM) into aerodigestive system. WTC associated morbidities include respiratory, gastrointestinal, chronic rhinosinusitis, cancer, mental health concerns and more recently a focus has been on cardiovascular disease. This proposal will investigate the development of WTC-cardiorespiratory and vascular dysfunction (WTC-CaRVD) which is firmly within the purview of the James Zadroga 9/11 Health and Compensation Act.

WTC-PM exposure causes heterogeneous obstructive airways disease (OAD) patterns, which include airway hyperreactivity (AHR) and loss of FEV1. Early diagnosis and therapeutic options are few, in part due to limited understanding of their pathogenesis. While pulmonary vascular changes are classically thought to occur due to the hypoxemia of late OAD, recent investigations show that vascular dysfunction occurs early in OAD. This vascular hypothesis of OAD postulates that pulmonary vasculature remodeling leads to loss of lung function. Early evidence of WTC-CaRVD includes increased prevalence of cardiovascular disease risk factors such as metabolic syndrome, elevated pulmonary artery/aorta ratio, and cardiovascular biomarkers (such as CRP). Murine models of WTC-PM exposure show inflammation, AHR both acutely and persistently and reflect what is seen in FDNY 1st responders. Airway and cardiac remodeling were also persistent features of WTC-PM exposure in the study team's murine models. Therefore, the study team will focus on Heme Oxygenase-1 (HO-1), a mediator of oxidative stress, known to stimulate collagen formation and is also induced after WTC-PM exposure. Furthermore, pathways and mechanisms of WTC-CaRVD warrant further study and are the focus of the 5-year proposal.

The HYPOTHESIS is that WTC-PM exposure causes WTC-CaRVD mediated by HO-1. First responders with AHR will have features of WTC-CaRVD, and will demonstrate a unique biomarker profile compared to controls.

ELIGIBILITY:
Inclusion Criteria:

1. Age 21-90
2. FDNY rescue and recovery worker
3. Documented WTC exposure
4. Consented/Enrolled member of the WTC-HP
5. Subjects are willing and able to consent for themselves to study enrollment
6. Subjects are willing and able to participate in study procedures
7. Are able to perform their activities of daily living independently
8. Are either light duty or retired FDNY Firefighters
9. Spirometry available within the last 24 months, and at a post-9/11 visit.
10. Have means to accommodate transportation to/from in-person visit Are able to attend a single visit at the CTSI (462 1st Avenue, C & D 4th Floor)
11. Pre-9/11 spirometry with FEV1%predicted ≥LLN and if not available 1st -post 9/11 spirometry with an FEV1 >80% predicted.
12. No recorded positive AHR testing prior to 9/11
13. Exposure at the WTC-site within 2 weeks of 9/11/2001
14. Entered WTC-HP before the site closure on 7/24/2002
15. Serum from their first post 9/11 WTC-HP visit is available in the biorepository and may be assayed
16. Are not currently being treated for malignancy
17. Subjects will either need to be defined as having WTC-AHR or be designated controls

Exclusion Criteria:

1. Unwilling to complete an informed consent.
2. Not enrolled in the WTC-HP
3. Do not meet eligibility criteria or did not have serum available in the biorepository from the first post 9/11 WTC-HP visit.
4. Have pre-existing and documented conditions or concurrent diagnoses, including (and not necessarily limited to) active cancer, severe heart disease, significant cognitive impairment, eating disorders, significant psychiatric illness, end-stage COPD, severe pulmonary hypertension, or organ transplant.
5. High dose steroid (>20mg prednisone or equivalent) or other hormonal treatments/chemotherapy use in the last month, including testosterone supplementation.
6. Life-expectancy < 6 months

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both Male and female subjects 21-90 year old will be enrolled. FDNY WTC exposed 1st responders enrolled in the WTC-Health Program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Levels of Heme Oxygenase-1 (HO-1) | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of Glutathione | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of Total Antioxidant Capacity (TAC) | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of Superoxide Dismutase (SOD) | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of Macrophage inflammatory protein-2 (MIP-2) | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of C-reactive protein (CRP) | up to Day 365
  All serum will be thawed once and assayed for biomarkers
Levels of fractional exhaled nitric oxide (FeNO) | up to Day 365
  FeNO will be quantified using NIOX VERO®
Score on St. George's Respiratory Questionnaire (SGRQ-C) | up to Day 365
  SGRQ-C is designed to assess how one's breathing is troubling a participant and how it affects one's life. The questionnaire consists of 14 questions. The total score range is 0-54; the higher the score, the worse the chest trouble.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Nolan, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Clinical & Translational Science Institute Clinical Research Center (CTSI CRC), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: The investigator who proposed to use the data and researchers who provide a methodologically sound proposal will have access to the data upon reasonable request. Requests should be directed to anna.nolan@med.nyu.edu. To gain access, data requestors will need to sign a data access agreement.